CLINICAL TRIAL: NCT04819113
Title: A PHASE 3B, OPEN-LABEL, STUDY TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF NIMENRIX(Registered) IN HEALTHY INFANTS, GIVEN AT 3 AND 12 MONTHS OF AGE
Brief Title: Study to Evaluate the Safety and Immunogenicity of Nimenrix (Registered) in Healthy Infants, Given at 3 and 12 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C0921062; 2020-005059-19 (EudraCT Number)
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Meningococcal Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimenrix (Experimental): Nimenrix
  Interventions: Biological: Nimenrix

INTERVENTIONS:
Biological: Nimenrix — MenACWY-TT vaccine

SUMMARY:
This study will evaluate the safety and immunogenicity of a single dose of Nimenrix in infants at 3 months of age, followed by a second dose at 12 months of age. Current posology allows for 2 doses of Nimenrix before 6 months of age, where the first dose is administered from 6 weeks onwards with a second dose at least 2 months later, with a booster at 12 months; and in infants from 6 months of age, a single dose at 6 months, with a booster dose at 12 months. This study will provide valuable immunogenicity and safety data for a single dose in healthy infants <6 months of age, followed by the booster at 12 months

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born at >36 weeks of gestation and who are 3 months of age (≥76 to ≤104 days) at the time of consent (the day of birth is considered day of life 1).
* Participants whose parent(s)/legal guardian(s) is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Healthy infants determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.
* Participants who are available for the duration of the study and whose parent(s)/legal guardian(s) can be contacted by telephone during study participation.
* Participants whose parent(s)/legal guardian(s) is capable of giving signed informed consent.

Exclusion Criteria:

* Previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* History of microbiologically proven disease caused by N meningitidis or Neisseria gonorrhoeae.
* Significant neurological disorder or history of seizure (including simple febrile seizure).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* Other medical or psychiatric condition, including recent or active suicidal ideation/behavior, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Major known congenital malformation or serious chronic disorder.
* Previous vaccination with any meningococcal vaccine containing groups A, C, W, or Y.

Ages: 76 Days to 104 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Finland (8):
  - Tampere Vaccine Research Clinic, Tampere, Pirkanmaa
  - Jarvenpaa Vaccine Research Center, Jarvenpaa, Uusimaa
  - Espoo Vaccine Research Clinic, Espoo
  - FVR, Etelä-Helsingin rokotetutkimusklinikka, Helsinki
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Jarvenpaa Vaccine Research Center, Jarvenpaa
  - Turku Vaccine Research Clinic, Turku
- Poland (5):
  - IN VIVO Bydgoszcz, Bydgoszcz
  - NZOZ Przychodnia Vitamed, Bydgoszcz
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow
  - GRAVITA. Diagnostyka i Leczenie nieplodnosci, Lodz
  - Szpital im. Św. Jadwigi Śląskiej w Trzebnicy, Trzebnica
- Spain (3):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruna
  - Hospital Universitario HM Sanchinarro, Madrid
  - Instituto Hispalense de Pediatria, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Koski S, Martinon-Torres F, Ramet M, Zolotas L, Newton R, Maansson R, Cutler M, Peyrani P, Findlow J, Balmer P, Jodar L, Gruber WC, Anderson AS, Beeslaar J. A Phase 3B, Open-Label Study to Evaluate the Immunogenicity and Safety of the Quadrivalent Meningococcal Nimenrix(R) Vaccine When Given to Healthy Infants at 3 and 12 Months of Age. Infect Dis Ther. 2025 Feb;14(2):463-481. doi: 10.1007/s40121-024-01098-8. Epub 2025 Jan 30. PMID 39883399
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0921062

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 153 participants were screened, of which 4 were screen failures.
Groups:
- Nimenrix: Participants aged 3 months were administered a single dose of 0.5 milliliter (mL) Nimenrix (Vaccination 1) intramuscularly into the left thigh muscle on Day 1 (Visit 1) and a second dose of Nimenrix (Vaccination 2) at 12 months of age (Visit 3). Participants had a safety follow-up visit 1 month after each vaccination (Visit 2 and Visit 4 respectively).
Period: Overall Study
Arm/Group | Nimenrix
Started | 149
Vaccination 1 | 147
Safety Population | 145
Vaccination 2 | 143
Completed | 143
Not Completed | 6
Not completed — Withdrawal by parent/guardian | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawn before vaccination | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 dose of investigational product and had safety data reported after vaccination.
Arm/Group | Nimenrix
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: Days] | 94.4 (6.09) [lower limit 6.09]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 141
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions included pain at injection site, redness and swelling and were recorded by the participant's parents/legal guardians in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: greater than (>) 0.0 to 2.0 cm; moderate: >2.0 to 7.0 cm; and severe: >7.0 cm. Pain at injection site was graded as mild: hurts if gently touched; moderate: hurts if gently touched with crying; severe: limited limb movement. Exact 2-sided confidence interval (CI) was based on the Clopper and Pearson method.
Time Frame: Within 7 days after vaccination 2
Population: Dose 2 safety population included participants who received the first and second dose of investigational product at Visit 1 and Visit 3 and for whom safety information was available from Visit 3. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 142
Percentage of participants
  Pain at injection site: Mild | 19.7 (13.5) [13.5 to 27.2]
  Pain at injection site: Moderate | 7.7 (3.9) [3.9 to 13.4]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 2.6]
  Redness: Mild | 14.1 (8.8) [8.8 to 20.9]
  Redness: Moderate | 2.8 (0.8) [0.8 to 7.1]
  Redness: Severe | 0 (0.0) [0.0 to 2.6]
  Swelling: Mild | 4.9 (2.0) [2.0 to 9.9]
  Swelling: Moderate | 1.4 (0.2) [0.2 to 5.0]
  Swelling: Severe | 0 (0.0) [0.0 to 2.6]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: Systemic events included fever, decreased appetite, increased sleep and irritability and were recorded by the participant's parents/legal guardians in an e-diary. Fever was defined as temperature greater than or equal to (>=) 38.0 degrees (deg) Celsius (C), categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C,>38.9 to 40.0 deg C and >40.0 deg C; decreased appetite graded as mild: decreased interest in eating, moderate: decreased oral intake and severe: refusal to feed; increased sleep graded as mild: increased or prolonged sleeping bouts, moderate: slightly subdued, interfered with daily activity and severe: disabling, not interested in usual daily activity; irritability graded as mild: easily consolable, moderate: required increased attention and severe: inconsolable, crying could not be comforted. Exact 2-sided CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 142
Percentage of participants
  Fever: >=38.0 deg C to 38.4 deg C | 6.3 (2.9) [2.9 to 11.7]
  Fever: >38.4 deg C to 38.9 deg C | 4.9 (2.0) [2.0 to 9.9]
  Fever: >38.9 deg C to 40.0 deg C | 3.5 (1.2) [1.2 to 8.0]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 2.6]
  Decreased appetite: Mild | 19.7 (13.5) [13.5 to 27.2]
  Decreased appetite: Moderate | 11.3 (6.6) [6.6 to 17.7]
  Decreased appetite: Severe | 1.4 (0.2) [0.2 to 5.0]
  Increased sleep: Mild | 38.0 (30.0) [30.0 to 46.5]
  Increased sleep: Moderate | 11.3 (6.6) [6.6 to 17.7]
  Increased sleep: Severe | 1.4 (0.2) [0.2 to 5.0]
  Irritability: Mild | 18.3 (12.3) [12.3 to 25.7]
  Irritability: Moderate | 42.3 (34.0) [34.0 to 50.8]
  Irritability: Severe | 2.8 (0.8) [0.8 to 7.1]

3. Primary Outcome: Percentage of Participants With Use of Antipyretic Medication Within 7 Days After Vaccination 2
Description: The use of antipyretic medication was recorded by the participant's parents/legal guardians in an e-diary for 7 days after vaccination. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 142
Percentage of participants | 55.6 (47.1) [47.1 to 64.0]

4. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 30 Days After Vaccination 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. Exact 2-sided CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Within 30 days after vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 143
Percentage of participants | 19.6 (13.4) [13.4 to 27.0]

5. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 30 Days After Vaccination 2
Description: An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 days after vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 143
Percentage of participants | 1.4 (0.2) [0.2 to 5.0]

6. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 30 Days After Vaccination 2
Description: An NDCMC was defined as a significant disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 days after vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 143
Percentage of participants | 0.0 (0.0) [0.0 to 2.5]

7. Primary Outcome: Percentage of Participants With Immediate AE Within 30 Minutes After Vaccination 2
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after administration of the investigational product. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 minutes after vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 143
Percentage of participants | 0.0 (0.0) [0.0 to 2.5]

8. Primary Outcome: Percentage of Participants Achieving Serum Bactericidal Assay Using Rabbit Complement (rSBA) Titers >=1:8 for Each Serogroup, Neisseria Meningitidis Group (Men) A, MenC, MenW-135 and MenY at Baseline: Post Dose 2 Evaluable Immunogenicity Population
Description: Percentage of participants achieving rSBA titer >=1:8 for each serogroup MenA, MenC, MenW-135 and MenY at baseline in participants who received vaccinations 1 and 2 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented. Analysis was performed on Post Dose (PD) 2 Evaluable Immunogenicity Population (EIP) (PD2 EIP).
Time Frame: At baseline (before vaccination 1)
Population: PD2 EIP: participants enrolled and eligible through 1 month after vaccination 2; received vaccine at visit (V) 1 and V3; blood drawn for assay testing within time frames at Month 0 (V1; before dose 1) and at 1 month after dose 2 (V4: window 28-42 days); at least 1 valid, determinate MenA, MenC, MenW-135, and MenY assay result at V4, received no prohibited vaccines/treatment and had no protocol deviations through V4. Here, N =participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 128
Percentage of participants
  MenA | 0.0 [0.0 to 2.8]
  MenC | 4.7 [1.7 to 9.9]
  MenW-135 | 0.8 [0.0 to 4.3]
  MenY | 7.8 [3.8 to 13.9]

9. Primary Outcome: Percentage of Participants Achieving rSBA Titers >= 1:8 for Each Serogroup MenA, MenC, MenW-135 and MenY at 1 Month After Vaccination 1: Post Dose 2 Evaluable Immunogenicity Population
Description: Percentage of participants achieving rSBA titer >=1:8 for each serogroup MenA, MenC, MenW-135 and MenY at 1 month after vaccination 1 in participants who received vaccination 1 and 2 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: 1 month after vaccination 1
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 124
Percentage of participants
  MenA | 82.3 [74.4 to 88.5]
  MenC | 91.1 [84.7 to 95.5]
  MenW-135 | 89.5 [82.7 to 94.3]
  MenY | 90.3 [83.7 to 94.9]

10. Primary Outcome: Percentage of Participants Achieving rSBA Titers >= 1:8 for Each Serogroup MenA, MenC, MenW-135 and MenY at Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: Percentage of participants achieving rSBA titer >=1:8 for each serogroup MenA, MenC, MenW-135 and MenY at vaccination 2 in participants who received vaccination 1 and 2 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: At vaccination 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 125
Percentage of participants
  MenA | 33.6 [25.4 to 42.6]
  MenC | 64.8 [55.8 to 73.1]
  MenW-135 | 67.2 [58.2 to 75.3]
  MenY | 66.4 [57.4 to 74.6]

11. Primary Outcome: Percentage of Participants Achieving rSBA Titers >= 1:8 for Each Serogroup MenA, MenC, MenW-135 and MenY at 1 Month After Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: Percentage of participants achieving rSBA titer >=1:8 for each serogroup MenA, MenC, MenW-135 and MenY at 1 month after vaccination 2 in participants who received vaccination 1 and 2 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: 1 month after vaccination 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 128
Percentage of participants
  MenA | 100.0 [97.2 to 100.0]
  MenC | 100.0 [97.2 to 100.0]
  MenW-135 | 100.0 [97.2 to 100.0]
  MenY | 100.0 [97.2 to 100.0]

12. Primary Outcome: Geometric Mean Titers (GMTs) of rSBA Titer for Each of MenA, MenC, MenW-135 and MenY Serogroups at Baseline: Post Dose 2 Evaluable Immunogenicity Population
Description: GMT was derived by calculating the mean on the natural log scale based on the t-distribution, then exponentiating the results. CIs were obtained by exponentiating the limits of CIs for the mean logarithm of the rSBA titers (based on the Student t distribution).
Time Frame: At baseline (before vaccination 1)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix
Number analyzed (Participants) | 128
Titer
  MenA | 4.0 [4.0 to 4.0]
  MenC | 4.4 [4.0 to 4.7]
  MenW-135 | 4.1 [3.9 to 4.3]
  MenY | 5.0 [4.3 to 5.8]

13. Primary Outcome: GMTs of rSBA Titer for Each of MenA, MenC, MenW-135 and MenY Serogroups at 1 Month After Vaccination 1: Post Dose 2 Evaluable Immunogenicity Population
Description: as for outcome 12
Time Frame: 1 month after vaccination 1
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix
Number analyzed (Participants) | 124
Titer
  MenA | 54.7 [41.1 to 72.9]
  MenC | 107.6 [81.3 to 142.5]
  MenW-135 | 202.4 [149.6 to 274.0]
  MenY | 187.2 [141.6 to 247.5]

14. Primary Outcome: GMTs of rSBA Titer for Each of MenA, MenC, MenW-135 and MenY Serogroups at Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: as for outcome 12
Time Frame: At vaccination 2
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix
Number analyzed (Participants) | 125
Titer
  MenA | 9.9 [7.6 to 13.0]
  MenC | 21.8 [16.1 to 29.5]
  MenW-135 | 21.7 [16.3 to 28.9]
  MenY | 24.5 [18.0 to 33.4]

15. Primary Outcome: GMTs of rSBA Titer for Each of MenA, MenC, MenW-135 and MenY Serogroups at 1 Month After Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: as for outcome 12
Time Frame: 1 month after vaccination 2
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix
Number analyzed (Participants) | 128
Titer
  MenA | 1818.0 [1497.8 to 2206.6]
  MenC | 1299.5 [1052.3 to 1604.9]
  MenW-135 | 2714.1 [2233.0 to 3298.8]
  MenY | 1667.1 [1393.9 to 1993.8]

16. Secondary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions included pain at injection site, redness and swelling and were recorded by the participant's parents/legal guardians in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: >0.0 to 2.0 cm; moderate: >2.0 to 7.0 cm; and severe: >7.0 cm. Pain at injection site was graded as mild: hurts if gently touched; moderate: hurts if gently touched with crying; severe: limited limb movement. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after vaccination 1
Population: Dose 1 safety population included participants who received the first dose of investigational product at Visit 1 and for whom safety information was available from Visit 1 to prior to Visit 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 145
Percentage of participants
  Pain at injection site: Mild | 13.8 (8.6) [8.6 to 20.5]
  Pain at injection site: Moderate | 2.8 (0.8) [0.8 to 6.9]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 2.5]
  Redness: Mild | 6.2 (2.9) [2.9 to 11.5]
  Redness: Moderate | 1.4 (0.2) [0.2 to 4.9]
  Redness: Severe | 0 (0.0) [0.0 to 2.5]
  Swelling: Mild | 1.4 (0.2) [0.2 to 4.9]
  Swelling: Moderate | 1.4 (0.2) [0.2 to 4.9]
  Swelling: Severe | 0 (0.0) [0.0 to 2.5]

17. Secondary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events included fever, decreased appetite, increased sleep and irritability and were recorded in e-diary. Fever was defined as temperature >=38.0 deg C, categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C,>38.9 to 40.0 deg C and >40.0 deg C; decreased appetite graded as mild: decreased interest in eating, moderate: decreased oral intake and severe: refusal to feed; increased sleep graded as mild: increased or prolonged sleeping bouts, moderate: slightly subdued, interfered with daily activity and severe: disabling, not interested in usual daily activity; irritability graded as mild: easily consolable, moderate: required increased attention and severe: inconsolable, crying could not be comforted. Exact 2-sided CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after vaccination 1
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 145
Percentage of participants
  Fever: >=38.0 deg C to 38.4 deg C | 7.6 (3.8) [3.8 to 13.2]
  Fever: >38.4 deg C to 38.9 deg C | 2.1 (0.4) [0.4 to 5.9]
  Fever: >38.9 deg C to 40.0 deg C | 0 (0.0) [0.0 to 2.5]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 2.5]
  Decreased appetite: Mild | 15.2 (9.8) [9.8 to 22.1]
  Decreased appetite: Moderate | 8.3 (4.3) [4.3 to 14.0]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 2.5]
  Increased sleep: Mild | 57.2 (48.8) [48.8 to 65.4]
  Increased sleep: Moderate | 7.6 (3.8) [3.8 to 13.2]
  Increased sleep: Severe | 1.4 (0.2) [0.2 to 4.9]
  Irritability: Mild | 27.6 (20.5) [20.5 to 35.6]
  Irritability: Moderate | 40.0 (32.0) [32.0 to 48.5]
  Irritability: Severe | 4.8 (2.0) [2.0 to 9.7]

18. Secondary Outcome: Percentage of Participants With Use of Antipyretic Medication Within 7 Days After Vaccination 1
Description: as for outcome 3
Time Frame: Within 7 days after vaccination 1
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 145
Percentage of participants | 39.3 (31.3) [31.3 to 47.8]

19. Secondary Outcome: Percentage of Participants With AEs Within 30 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. Exact 2-sided CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Within 30 days after vaccination 1
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 145
Percentage of participants | 6.9 (3.4) [3.4 to 12.3]

20. Secondary Outcome: Percentage of Participants With SAEs and NDCMCs: Within 30 Days After Vaccination 1, From 1 Month After Vaccination 1 to 9 Months After Vaccination 1, From Vaccination 1 to 9 Months After Vaccination 1
Description: An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. An NDCMC was defined as a significant disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 days after vaccination 1, from 1 month after vaccination 1 to 9 months after vaccination 1 and from vaccination 1 to 9 months after vaccination 1
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 145
Percentage of participants
  SAE: Within 30 days after Vaccination 1 | 1.4 [0.2 to 4.9]
  SAE: From 1 Month after Vaccination 1 to 9 Month after Vaccination 1 | 4.1 [1.5 to 8.8]
  SAE: From Vaccination 1 to 9 Month after Vaccination 1 | 5.5 [2.4 to 10.6]
  NDCMC: Within 30 days after Vaccination 1 | 0.0 [0.0 to 2.5]
  NDCMC:From 1 Month after Vaccination 1 to 9 Month after Vaccination 1 | 0.0 [0.0 to 2.5]
  NDCMC: From Vaccination 1 to 9 Month after Vaccination 1 | 0.0 [0.0 to 2.5]

21. Secondary Outcome: Percentage of Participants With Immediate AE Within 30 Minutes After Vaccination 1
Description: as for outcome 7
Time Frame: Within 30 minutes after vaccination 1
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 145
Percentage of participants | 0.0 (0.0) [0.0 to 2.5]

22. Secondary Outcome: Percentage of Participants Achieving rSBA Titers >= 1:8 for Each Serogroup MenA, MenC, MenW-135 and MenY at Baseline and 1 Month After Vaccination 1: Post Dose 1 Evaluable Immunogenicity Population
Description: Percentage of participants achieving rSBA titer >=1:8 for each serogroup MenA, MenC, MenW-135 and MenY at baseline and 1 month after Vaccination 1 in participants who received Vaccination 1 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented. Analysis was performed on post-dose 1 (PD1) evaluable immunogenicity population (EIP).
Time Frame: At baseline (before vaccination 1) and 1 month after vaccination 1
Population: PD1 EIP: participants enrolled and eligible through V2; received vaccine at V1; blood drawn for assay testing within time frames at Month 0 (V1; before dose 1) and Month 1 (V2; 1 month after dose 1: window 28-42 days); had at least 1 valid, determinate MenA, MenC, MenW-135 and MenY assay result at V2, received no prohibited vaccines/treatment and had no protocol deviations through V2. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 116
Percentage of participants
  MenA, Baseline (Before Vaccination 1) | 0.0 [0.0 to 3.1]
  MenA, 1 Month after Vaccination 1 | 81.0 [72.7 to 87.7]
  MenC, Baseline (Before Vaccination 1) | 5.2 [1.9 to 10.9]
  MenC, 1 Month after Vaccination 1 | 89.7 [82.6 to 94.5]
  MenW-135, Baseline (Before Vaccination 1) | 0.9 [0.0 to 4.7]
  MenW-135, 1 Month after Vaccination 1 | 88.8 [81.6 to 93.9]
  MenY, Baseline (Before Vaccination 1) | 7.8 [3.6 to 14.2]
  MenY, 1 Month after Vaccination 1 | 87.9 [80.6 to 93.2]

23. Secondary Outcome: Percentage of Participants Achieving rSBA Titers >= 1:128 for Each Serogroup MenA, MenC, MenW-135 and MenY at Baseline and 1 Month After Vaccination 1: Post Dose 1 Evaluable Immunogenicity Population
Description: Percentage of participants achieving rSBA titer >= 1:128 for each serogroup MenA, MenC, MenW-135 and MenY at baseline and 1 month after vaccination 1 in participants who received vaccination 1 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: At baseline (before vaccination 1) and 1 month after vaccination 1
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 116
Percentage of participants
  MenA, Baseline (Before Vaccination 1) | 0.0 [0.0 to 3.1]
  MenA, 1 Month after Vaccination 1 | 35.3 [26.7 to 44.8]
  MenC, Baseline (Before Vaccination 1) | 0.0 [0.0 to 3.1]
  MenC, 1 Month after Vaccination 1 | 65.5 [56.1 to 74.1]
  MenW-135, Baseline (Before Vaccination 1) | 0.9 [0.0 to 4.7]
  MenW-135, 1 Month after Vaccination 1 | 79.3 [70.8 to 86.3]
  MenY, Baseline (Before Vaccination 1) | 2.6 [0.5 to 7.4]
  MenY, 1 Month after Vaccination 1 | 81.0 [72.7 to 87.7]

24. Secondary Outcome: GMTs of rSBA Titer for Each of MenA, MenC, MenW-135 and MenY Serogroups at Baseline and 1 Month After Vaccination 1: Post Dose 1 Evaluable Immunogenicity Population
Description: as for outcome 12
Time Frame: At baseline (before vaccination 1) and 1 month after vaccination 1
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix
Number analyzed (Participants) | 116
Titer
  MenA, Baseline (Before Vaccination 1) | 4.0 [4.0 to 4.0]
  MenA, 1 Month after Vaccination 1 | 50.1 [37.2 to 67.5]
  MenC, Baseline (Before Vaccination 1) | 4.3 [4.0 to 4.5]
  MenC, 1 Month after Vaccination 1 | 96.7 [71.8 to 130.1]
  MenW-135, Baseline (Before Vaccination 1) | 4.1 [3.9 to 4.4]
  MenW-135, 1 Month after Vaccination 1 | 193.3 [140.8 to 265.5]
  MenY, Baseline (Before Vaccination 1) | 4.8 [4.2 to 5.4]
  MenY, 1 Month after Vaccination 1 | 172.6 [126.6 to 235.2]

25. Secondary Outcome: Percentage of Participants Achieving Serum Bactericidal Assay Using Human Complement (hSBA) Titers >= 1:4 for Each Serogroup MenA, MenC, MenW-135 and MenY at Baseline and 1 Month After Vaccination 1: Post Dose 1 Evaluable Immunogenicity Population
Description: Percentage of participants achieving hSBA titers >= 1:4 for each serogroup MenA, MenC, MenW-135 and MenY at baseline and 1 month after vaccination 1 in participants who received Vaccination 1 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: At baseline (before vaccination 1) and 1 month after vaccination 1
Population: PD1 EIP:participants enrolled & eligible through V2;received vaccine at V1;blood drawn for assay testing within time frames at Month 0 (V1; before dose1) & Month1 (V2;1 month after dose1:window 28-42 days); had at least 1 valid, determinate MenA, MenC, MenW-135 & MenY assay result at V2, received no prohibited vaccines/treatment & had no protocol deviation through V2.N=signifies participants evaluable for this outcome measure.'Number Analyzed' signifies participants evaluable for specified row
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 107
Percentage of participants
  MenA, Baseline (Before Vaccination 1): number analyzed (Participants) | 92
  MenA, Baseline (Before Vaccination 1) | 7.6 [3.1 to 15.1]
  MenA, 1 Month after Vaccination 1: number analyzed (Participants) | 106
  MenA, 1 Month after Vaccination 1 | 94.3 [88.1 to 97.9]
  MenC, Baseline (Before Vaccination 1): number analyzed (Participants) | 100
  MenC, Baseline (Before Vaccination 1) | 13.0 [7.1 to 21.2]
  MenC, 1 Month after Vaccination 1 | 91.6 [84.6 to 96.1]
  MenW-135, Baseline (Before Vaccination 1): number analyzed (Participants) | 58
  MenW-135, Baseline (Before Vaccination 1) | 13.8 [6.1 to 25.4]
  MenW-135, 1 Month after Vaccination 1: number analyzed (Participants) | 62
  MenW-135, 1 Month after Vaccination 1 | 33.9 [22.3 to 47.0]
  MenY, Baseline (Before Vaccination 1): number analyzed (Participants) | 66
  MenY, Baseline (Before Vaccination 1) | 25.8 [15.8 to 38.0]
  MenY, 1 Month after Vaccination 1: number analyzed (Participants) | 68
  MenY, 1 Month after Vaccination 1 | 48.5 [36.2 to 61.0]

26. Secondary Outcome: Percentage of Participants Achieving hSBA Titers >= 1:8 for Each Serogroup MenA, MenC, MenW-135 and MenY at Baseline and 1 Month After Vaccination 1: Post Dose 1 Evaluable Immunogenicity Population
Description: Percentage of participants achieving hSBA titers >= 1:8 for each serogroup MenA, MenC, MenW-135 and MenY at baseline and 1 month after vaccination 1 in participants who received Vaccination 1 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: At baseline (before vaccination 1) and 1 month after vaccination 1
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 107
Percentage of participants
  MenA, Baseline (Before Vaccination 1): number analyzed (Participants) | 92
  MenA, Baseline (Before Vaccination 1) | 6.5 [2.4 to 13.7]
  MenA, 1 Month after Vaccination 1: number analyzed (Participants) | 106
  MenA, 1 Month after Vaccination 1 | 94.3 [88.1 to 97.9]
  MenC, Baseline (Before Vaccination 1): number analyzed (Participants) | 100
  MenC, Baseline (Before Vaccination 1) | 13.0 [7.1 to 21.2]
  MenC, 1 Month after Vaccination 1 | 91.6 [84.6 to 96.1]
  MenW-135, Baseline (Before Vaccination 1): number analyzed (Participants) | 58
  MenW-135, Baseline (Before Vaccination 1) | 13.8 [6.1 to 25.4]
  MenW-135, 1 Month after Vaccination 1: number analyzed (Participants) | 62
  MenW-135, 1 Month after Vaccination 1 | 33.9 [22.3 to 47.0]
  MenY, Baseline (Before Vaccination 1): number analyzed (Participants) | 66
  MenY, Baseline (Before Vaccination 1) | 25.8 [15.8 to 38.0]
  MenY, 1 Month after Vaccination 1: number analyzed (Participants) | 68
  MenY, 1 Month after Vaccination 1 | 48.5 [36.2 to 61.0]

27. Secondary Outcome: GMTs of hSBA Titer for Each of MenA, MenC, MenW-135 and MenY Serogroups at Baseline and 1 Month After Vaccination 1: Post Dose 1 Evaluable Immunogenicity Population
Description: GMT was derived by calculating the mean on the natural log scale based on the t-distribution, then exponentiating the results. CIs were obtained by exponentiating the limits of CIs for the mean logarithm of the hSBA titers (based on the Student t distribution).
Time Frame: At baseline (before vaccination 1) and 1 month after vaccination 1
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix
Number analyzed (Participants) | 107
Titer
  MenA, Baseline (Before Vaccination 1): number analyzed (Participants) | 92
  MenA, Baseline (Before Vaccination 1) | 2.4 [2.1 to 2.7]
  MenA, 1 Month after Vaccination 1: number analyzed (Participants) | 106
  MenA, 1 Month after Vaccination 1 | 82.0 [63.9 to 105.0]
  MenC, Baseline (Before Vaccination 1): number analyzed (Participants) | 100
  MenC, Baseline (Before Vaccination 1) | 2.9 [2.4 to 3.6]
  MenC, 1 Month after Vaccination 1 | 128.4 [93.3 to 176.8]
  MenW-135, Baseline (Before Vaccination 1): number analyzed (Participants) | 58
  MenW-135, Baseline (Before Vaccination 1) | 2.9 [2.3 to 3.7]
  MenW-135, 1 Month after Vaccination 1: number analyzed (Participants) | 62
  MenW-135, 1 Month after Vaccination 1 | 6.9 [4.4 to 10.9]
  MenY, Baseline (Before Vaccination 1): number analyzed (Participants) | 66
  MenY, Baseline (Before Vaccination 1) | 6.6 [3.9 to 11.3]
  MenY, 1 Month after Vaccination 1: number analyzed (Participants) | 68
  MenY, 1 Month after Vaccination 1 | 19.2 [10.2 to 36.3]

28. Secondary Outcome: Percentage of Participants Achieving hSBA Titers >= 1:4 for Each Serogroup MenA, MenC, MenW-135 and MenY at Baseline, 1 Month After Vaccination 1, at Vaccination 2 and 1 Month After Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: Percentage of participants achieving hSBA titers >= 1:4 for each serogroup MenA, MenC, MenW-135 and MenY at baseline, 1 month after vaccination 1, at vaccination 2 and 1 month after vaccination 2 in participants who received vaccination 1 and 2 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: At baseline (before vaccination 1), 1 month after vaccination 1, at vaccination 2 and 1 month after vaccination 2
Population: PD2 EIP:participant enrolled & eligible through 1month after vaccination2;received vaccine at V1 &V3;blood drawn for assay testing within time frame at Month0 (V1;before dose1) & at 1 month after dose2 (V4:window 28-42 days); at least 1 valid, determinate MenA, MenC, MenW-135, & MenY assay result at V4, received no prohibited vaccine/treatment & had no protocol deviation through V4.Here,N=participant evaluable for outcome measure.'Number Analyzed' signify participant evaluable for specified row
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 123
Percentage of participants
  MenA, Baseline (Before Vaccination 1): number analyzed (Participants) | 100
  MenA, Baseline (Before Vaccination 1) | 8.0 [3.5 to 15.2]
  MenA, 1 Month after Vaccination 1: number analyzed (Participants) | 111
  MenA, 1 Month after Vaccination 1 | 95.5 [89.8 to 98.5]
  MenA, Before Vaccination 2: number analyzed (Participants) | 108
  MenA, Before Vaccination 2 | 49.1 [39.3 to 58.9]
  MenA, 1 Month after Vaccination 2 | 100.0 [97.0 to 100.0]
  MenC, Baseline (Before Vaccination 1): number analyzed (Participants) | 111
  MenC, Baseline (Before Vaccination 1) | 11.7 [6.4 to 19.2]
  MenC, 1 Month after Vaccination 1: number analyzed (Participants) | 116
  MenC, 1 Month after Vaccination 1 | 93.1 [86.9 to 97.0]
  MenC, Before Vaccination 2: number analyzed (Participants) | 121
  MenC, Before Vaccination 2 | 85.1 [77.5 to 90.9]
  MenC, 1 Month after Vaccination 2 | 100.0 [97.0 to 100.0]
  MenW-135, Baseline (Before Vaccination 1): number analyzed (Participants) | 65
  MenW-135, Baseline (Before Vaccination 1) | 12.3 [5.5 to 22.8]
  MenW-135, 1 Month after Vaccination 1: number analyzed (Participants) | 67
  MenW-135, 1 Month after Vaccination 1 | 38.8 [27.1 to 51.5]
  MenW-135, Before Vaccination 2: number analyzed (Participants) | 100
  MenW-135, Before Vaccination 2 | 94.0 [87.4 to 97.8]
  MenW-135, 1 Month after Vaccination 2: number analyzed (Participants) | 119
  MenW-135, 1 Month after Vaccination 2 | 100.0 [96.9 to 100.0]
  MenY, Baseline (Before Vaccination 1): number analyzed (Participants) | 73
  MenY, Baseline (Before Vaccination 1) | 21.9 [13.1 to 33.1]
  MenY, 1 Month after Vaccination 1: number analyzed (Participants) | 72
  MenY, 1 Month after Vaccination 1 | 50.0 [38.0 to 62.0]
  MenY, Before Vaccination 2: number analyzed (Participants) | 106
  MenY, Before Vaccination 2 | 70.8 [61.1 to 79.2]
  MenY, 1 Month after Vaccination 2 | 100.0 [97.0 to 100.0]

29. Secondary Outcome: Percentage of Participants Achieving hSBA Titers >= 1:8 for Each Serogroup MenA, MenC, MenW-135 and MenY at Baseline, 1 Month After Vaccination 1, at Vaccination 2 and 1 Month After Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: Percentage of participants achieving hSBA titers >= 1:8 for each serogroup MenA, MenC, MenW-135 and MenY at baseline, 1 month after vaccination 1, at vaccination 2 and 1 month after vaccination 2 in participants who received vaccination 1 and 2 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: At baseline (before vaccination 1), 1 month after vaccination 1, at vaccination 2 and 1 month after vaccination 2
Population: PD2 EIP:participant enrolled & eligible through 1month after vaccination2;received vaccine at visit 1,3;blood drawn for assay testing within time frames at Month0 (V1;before dose1) & at 1month after dose2(V4:window 28-42 days);at least 1 valid,determinate MenA, MenC,MenW-135, & MenY assay result at V4,received no prohibited vaccine/treatment & had no protocol deviation through V4.Here,N=participant evaluable for outcome measure. 'Number Analyzed' signify participant evaluable for specified row.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 123
Percentage of participants
  MenA, Baseline (Before Vaccination 1): number analyzed (Participants) | 100
  MenA, Baseline (Before Vaccination 1) | 7.0 [2.9 to 13.9]
  MenA, 1 Month after Vaccination 1: number analyzed (Participants) | 111
  MenA, 1 Month after Vaccination 1 | 95.5 [89.8 to 98.5]
  MenA, Baseline (Before Vaccination 2): number analyzed (Participants) | 108
  MenA, Baseline (Before Vaccination 2) | 46.3 [36.7 to 56.2]
  MenA, 1 Month after Vaccination 2 | 100.0 [97.0 to 100.0]
  MenC, Baseline (Before Vaccination 1): number analyzed (Participants) | 111
  MenC, Baseline (Before Vaccination 1) | 11.7 [6.4 to 19.2]
  MenC, 1 Month after Vaccination 1: number analyzed (Participants) | 116
  MenC, 1 Month after Vaccination 1 | 93.1 [86.9 to 97.0]
  MenC, Baseline (Before Vaccination 2): number analyzed (Participants) | 121
  MenC, Baseline (Before Vaccination 2) | 85.1 [77.5 to 90.9]
  MenC, 1 Month after Vaccination 2 | 100.0 [97.0 to 100.0]
  MenW-135, Baseline (Before Vaccination 1): number analyzed (Participants) | 65
  MenW-135, Baseline (Before Vaccination 1) | 12.3 [5.5 to 22.8]
  MenW-135, 1 Month after Vaccination 1: number analyzed (Participants) | 67
  MenW-135, 1 Month after Vaccination 1 | 38.8 [27.1 to 51.5]
  MenW-135, Baseline (Before Vaccination 2): number analyzed (Participants) | 100
  MenW-135, Baseline (Before Vaccination 2) | 94.0 [87.4 to 97.8]
  MenW-135, 1 Month after Vaccination 2: number analyzed (Participants) | 119
  MenW-135, 1 Month after Vaccination 2 | 100.0 [96.9 to 100.0]
  MenY, Baseline (Before Vaccination 1): number analyzed (Participants) | 73
  MenY, Baseline (Before Vaccination 1) | 21.9 [13.1 to 33.1]
  MenY, 1 Month after Vaccination 1: number analyzed (Participants) | 72
  MenY, 1 Month after Vaccination 1 | 50.0 [38.0 to 62.0]
  MenY, Baseline (Before Vaccination 2): number analyzed (Participants) | 106
  MenY, Baseline (Before Vaccination 2) | 70.8 [61.1 to 79.2]
  MenY, 1 Month after Vaccination 2 | 100.0 [97.0 to 100.0]

30. Secondary Outcome: GMTs of hSBA Titer for Each of MenA, MenC, MenW-135 and MenY Serogroups at Baseline, 1 Month After Vaccination 1, at Vaccination 2 and 1 Month After Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: as for outcome 27
Time Frame: At baseline (before vaccination 1), 1 month after vaccination 1, at vaccination 2 and 1 month after vaccination 2
Population: PD2 EIP:participants enrolled & eligible through 1 month after vaccination2; received vaccine at visit (V) 1 & V3;blood drawn for assay testing within time frames at Month0 (V1; before dose 1) & at 1 month after dose2 (V4: window 28-42 days);at least 1 valid,determinate MenA, MenC, MenW-135, & MenY assay result at V4,received no prohibited vaccines/treatment & had no protocol deviation through V4.Here,N=participants evaluable for this outcome measure & n=participant evaluable for specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix
Number analyzed (Participants) | 123
Titer
  MenA, Baseline (Before Vaccination 1): number analyzed (Participants) | 100
  MenA, Baseline (Before Vaccination 1) | 2.4 [2.1 to 2.7]
  MenA, 1 Month after Vaccination 1: number analyzed (Participants) | 111
  MenA, 1 Month after Vaccination 1 | 86.9 [68.8 to 109.8]
  MenA, Baseline (Before Vaccination 2): number analyzed (Participants) | 108
  MenA, Baseline (Before Vaccination 2) | 9.5 [6.8 to 13.2]
  MenA, 1 Month after Vaccination 2 | 1208.4 [976.9 to 1494.8]
  MenC, Baseline (Before Vaccination 1): number analyzed (Participants) | 111
  MenC, Baseline (Before Vaccination 1) | 2.9 [2.3 to 3.6]
  MenC, 1 Month after Vaccination 1: number analyzed (Participants) | 116
  MenC, 1 Month after Vaccination 1 | 149.8 [111.3 to 201.6]
  MenC, Baseline (Before Vaccination 2): number analyzed (Participants) | 121
  MenC, Baseline (Before Vaccination 2) | 74.8 [52.3 to 107.0]
  MenC, 1 Month after Vaccination 2 | 7299.6 [5362.8 to 9936.0]
  MenW-135, Baseline (Before Vaccination 1): number analyzed (Participants) | 65
  MenW-135, Baseline (Before Vaccination 1) | 2.8 [2.2 to 3.5]
  MenW-135, 1 Month after Vaccination 1: number analyzed (Participants) | 67
  MenW-135, 1 Month after Vaccination 1 | 8.8 [5.5 to 14.2]
  MenW-135, Baseline (Before Vaccination 2): number analyzed (Participants) | 100
  MenW-135, Baseline (Before Vaccination 2) | 121.6 [90.0 to 164.2]
  MenW-135, 1 Month after Vaccination 2: number analyzed (Participants) | 119
  MenW-135, 1 Month after Vaccination 2 | 6955.8 [5922.4 to 8169.4]
  MenY, Baseline (Before Vaccination 1): number analyzed (Participants) | 73
  MenY, Baseline (Before Vaccination 1) | 5.7 [3.5 to 9.5]
  MenY, 1 Month after Vaccination 1: number analyzed (Participants) | 72
  MenY, 1 Month after Vaccination 1 | 19.9 [10.8 to 36.6]
  MenY, Baseline (Before Vaccination 2): number analyzed (Participants) | 106
  MenY, Baseline (Before Vaccination 2) | 45.7 [28.8 to 72.5]
  MenY, 1 Month after Vaccination 2 | 5062.1 [4202.9 to 6097.0]

31. Secondary Outcome: Percentage of Participants Achieving rSBA Titers >= 1:128 for Each Serogroup MenA, MenC, MenW-135 and MenY at Baseline, 1 Month After Vaccination 1, at Vaccination 2 and 1 Month After Vaccination 2: Post Dose 2 Evaluable Immunogenicity Population
Description: Percentage of participants achieving rSBA Titers >= 1:128 for each serogroup MenA, MenC, MenW-135 and MenY at baseline, 1 month after vaccination 1, at vaccination 2 and 1 month after vaccination 2 in Participants who received vaccination 1 and 2 were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: At baseline (before vaccination 1), 1 month after vaccination 1, at vaccination 2 and 1 month after vaccination 2
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nimenrix
Number analyzed (Participants) | 128
Percentage of participants
  MenA, Baseline (Before Vaccination 1) | 0 [0.0 to 2.8]
  MenA, 1 Month after Vaccination 1: number analyzed (Participants) | 124
  MenA, 1 Month after Vaccination 1 | 40.3 [31.6 to 49.5]
  MenA, Before Vaccination 2: number analyzed (Participants) | 125
  MenA, Before Vaccination 2 | 15.2 [9.4 to 22.7]
  MenA, 1 Month after Vaccination 2 | 100.0 [97.2 to 100.0]
  MenC, Baseline (Before Vaccination 1) | 0.8 [0.0 to 4.3]
  MenC, 1 Month after Vaccination 1: number analyzed (Participants) | 124
  MenC, 1 Month after Vaccination 1 | 67.7 [58.8 to 75.9]
  MenC, Before Vaccination 2: number analyzed (Participants) | 125
  MenC, Before Vaccination 2 | 20.8 [14.1 to 29.0]
  MenC, 1 Month after Vaccination 2 | 98.4 [94.5 to 99.8]
  MenW-135, Baseline (Before Vaccination 1) | 0.8 [0.0 to 4.3]
  MenW-135, 1 Month after Vaccination 1: number analyzed (Participants) | 124
  MenW-135, 1 Month after Vaccination 1 | 79.8 [71.7 to 86.5]
  MenW-135, Before Vaccination 2: number analyzed (Participants) | 125
  MenW-135, Before Vaccination 2 | 23.2 [16.1 to 31.6]
  MenW-135, 1 Month after Vaccination 2 | 100.0 [97.2 to 100.0]
  MenY, Baseline (Before Vaccination 1) | 3.9 [1.3 to 8.9]
  MenY, 1 Month after Vaccination 1: number analyzed (Participants) | 124
  MenY, 1 Month after Vaccination 1 | 83.1 [75.3 to 89.2]
  MenY, Before Vaccination 2: number analyzed (Participants) | 125
  MenY, Before Vaccination 2 | 27.2 [19.6 to 35.9]
  MenY, 1 Month after Vaccination 2 | 99.2 [95.7 to 100.0]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events were recorded using systematic assessment within 7 days after Vaccination 1 and 2; SAEs and all-cause mortality recorded using non-systematic assessment from Day 1 up to 42 days after Vaccination 2 (approximately 10 months and 12 days); other AEs recorded using non-systematic assessment from Day 1 up to 42 days after Vaccination 1 and from Day of Vaccination 2 up to 42 days after Vaccination 2
Description: Same event may appear as both an SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population included all enrolled participants who received at least 1 dose of investigational product and had safety data reported after vaccination.
Arm/Group | Nimenrix
All-Cause Mortality (participants affected / at risk) | 0/145
Serious Adverse Events (participants affected / at risk) | 10/145
Other Adverse Events (participants affected / at risk) | 139/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix (N=145)
Food protein-induced enterocolitis syndrome (Gastrointestinal disorders) | 1
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3
Respiratory syncytial virus infection (Infections and infestations) | 2
Concussion (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix (N=145)
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 51
Pyrexia (General disorders) | 5
Pyrexia (FEVER) (General disorders) | 31
Swelling (SWELLING) (General disorders) | 12
Bronchiolitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Hand-foot-and-mouth disease (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 8
Otitis media (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 7
Viral infection (Infections and infestations) | 2
Head injury (Injury, poisoning and procedural complications) | 2
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 65
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 115
Irritability (IRRITABILITY) (Psychiatric disorders) | 119
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04819113/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT04819113/SAP_001.pdf